CLINICAL TRIAL: NCT03839693
Title: Clinical Trial to Evaluate ET-01 in Subjects With Lateral Canthal Lines
Brief Title: ET-01 in Subjects With Lateral Canthal Lines, LCL-208
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eirion Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ET-01-LCL-208
Record Dates: First submitted 2019-02-08; First posted 2019-02-15 (Actual); Results first posted 2022-07-26 (Actual); Last update posted 2022-08-23 (Actual); Status verified 2022-07

CONDITIONS: Lateral Canthal Lines; Crow's Feet
MeSH Terms: interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Intervention Model Description: sequential cohort, dose escalating study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Vehicle (Placebo Comparator): Vehicle
  Interventions: Biological: Vehicle
- ET-01 345U (Experimental): botulinum toxin, Type A, Dose 1, 345 U
  Interventions: Biological: botulinum toxin, Type A
- ET-01 1100U (Experimental): botulinum toxin, Type A, Dose 2, 1100 U
  Interventions: Biological: botulinum toxin, Type A

INTERVENTIONS:
Biological: botulinum toxin, Type A — topical liniment
  Other Names: ET-01
  Arms: ET-01 1100U; ET-01 345U
Biological: Vehicle — Vehicle Formulation
  Arms: Vehicle

SUMMARY:
This study tests an investigational drug formulation called ET-01, botulinum toxin, Type A, topical, in lateral canthal lines (LCL).

DETAILED DESCRIPTION:
This product is being tested for its ability to reduce lateral canthal lines, also known as Crow's Feet.

ELIGIBILITY:
Inclusion Criteria:

* females 25 - 65 years of age
* minimal to moderate Crow's Feet wrinkles at rest
* moderate to severe Crow's Feet on contraction
* adequate vision to assess facial wrinkles in a mirror
* willingness to refrain from products affecting skin remodeling
* female subjects must be not pregnant and non-lactating
* subjects should be in good general health

Exclusion Criteria:

* history of adverse reactions to any prior botulinum toxin treatments
* history of vaccination or non-response to any prior botulinum toxin treatments
* botulinum toxin treatment in the prior 6 months
* present or history of neuromuscular disease, eyelid ptosis, muscle weakness, paralysis, or "dry eye"
* history of peri-ocular surgery, brow lift or related procedures
* procedures affecting the lateral canthal region in the prior 12 months
* application of topical prescription medication to the treatment area
* female subjects who are pregnant or are nursing a child

Ages: 25 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2018-10-16 (Actual); Primary Completion 2019-04-18 (Actual); Study Completion 2019-09-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Baumann Cosmetic & Research Institute, Miami, Florida
  - Synexus, Inc., Pinellas Park, Florida
  - Forefront Dermatology, Louisville, Kentucky
  - Westlake Dermatology Clinical Research Center, Austin, Texas
  - Virginia Clinical Research, Inc., Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from five medical centers between October 2018 and March 2019.
Pre-assignment Details: A total of N=88 subjects were screened; N=75 were found eligible and were randomized and treated.
Groups:
- ET-01 345U: botulinum toxin, Type A, Dose 1, 345U
  lower dose of botulinum toxin, Type A: topical liniment
- ET-01 1100U: botulinum toxin, Type A, Dose 2, 1100U
  higher dose of botulinum toxin, Type A: topical liniment
Period: Overall Study
Arm/Group | Vehicle | ET-01 345U | ET-01 1100U
Started | 25 | 30 | 20
Completed | 23 | 28 | 16
Not Completed | 2 | 2 | 4
Not completed — Lost to Follow-up | 0 | 2 | 2
Not completed — Withdrawal by Subject | 1 | 0 | 2
Not completed — subject moved out of the area | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- ET-01 345U: botulinum toxin, Type A, Lower Dose 1, 345U
  botulinum toxin, Type A: topical liniment
- ET-01 1100U: botulinum toxin, Type A, Higher Dose 2, 1100U
  botulinum toxin, Type A: topical liniment
- Total: Total of all reporting groups
Arm/Group | Vehicle | ET-01 345U | ET-01 1100U | Total
Number analyzed (Participants) | 25 | 30 | 20 | 75
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 23 | 29 | 19 | 71
  >=65 years | 2 | 1 | 1 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 30 | 20 | 75
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 4 | 6 | 12
  Not Hispanic or Latino | 22 | 25 | 14 | 61
  Unknown or Not Reported | 1 | 1 | 0 | 2
IGA-C [Mean (Standard Deviation); unit: units on a scale] — Investigator Global Assessment on Contraction using the ordinal Crow's Feet Wrinkle Scale where severity is scored between 0=absent and 4=severe.
  units on a scale | 3.3 (0.4) | 3.5 (0.5) | 3.5 (0.5) | 3.4 (0.5)
SSA-C [Mean (Standard Deviation); unit: units on a scale] — Subject Self-Assessment. Crow's Feet Wrinkle Scale where severity is scored between 0-4 (0=absent; 4=severe).
  units on a scale | 3.5 (0.5) | 3.7 (0.5) | 3.8 (0.4) | 3.6 (0.5)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Response Defined as Change in IGA-C (Investigators Global Assessment) Score by at Least 2 Ordinals From Baseline to Week 4
Description: Investigators Global Assessment of the Crow's Feet Wrinkle Scale where severity is scored between 0-4 (0=absent; 4=severe). Response is defined as change by at least two ordinals from Baseline to Week 4.
Time Frame: Week 4
Population: Intent-To-Treat (ITT) population defined as all treated subjects who had at least one post-baseline visit. No imputation was performed when only incomplete data were available.
Measure: Count of Participants; unit: Participants
Groups:
- ET-01 345U: botulinum toxin, Type A, Dose 1
  botulinum toxin, Type A: topical liniment
- ET-01 1100U: botulinum toxin, Type A, Dose 2
  botulinum toxin, Type A: topical liniment
Arm/Group | Vehicle | ET-01 345U | ET-01 1100U
Number analyzed (Participants) | 23 | 30 | 19
Participants | 2 | 0 | 1

2. Secondary Outcome: Total Number of Observations With a Response Defined as Change ≥2 in IGA-C and SSA-C Score at Any Post Baseline Visit
Description: Total number of observations with a change in the Investigators Global Assessment on Contraction, IGA-C, and the Subject Self-Assessment on Contraction, SSA-C, using the Crow's Feet Wrinkle Scale, where severity is scored between 0-4 (0=absent; 4=severe). To count, a "responder" is defined as a change by at least two ordinals in both assessments. The observation period includes all post-baseline visits from Week 1 to Week 26.
Time Frame: Week 1, 2, 4, 8,12,18, and 26
Population: as for outcome 1
Measure: Count of Units; unit: Observations
Units Other Than Participants: Observations
Arm/Group | Vehicle | ET-01 345U | ET-01 1100U
Number analyzed (Participants) | 25 | 30 | 20
Number analyzed (Observations) | 162 | 202 | 131
Observations | 1 | 5 | 5

3. Secondary Outcome: Total Number of Observations With a Response Defined as Change in SSA-C Score ≥ 2 at Any Time Between Week 4 and Week 12
Description: Total number of observations with a change by at least two ordinals in the Subjects Self-Assessment on Contraction, SSA-C, using the Crow's Feet Wrinkle Scale, where severity is scored between 0-4 (0=absent; 4=severe). To count, a "responder" is defined as an improvement ≥ 2 score points. The observation period covers the time time of expected peak efficacy from Week 4 to Week 12.
Time Frame: Week 4, 8,and 12
Population: as for outcome 1
Measure: Count of Units; unit: Observations
Units Other Than Participants: Observations
Groups:
- ET-01 345U: botulinum toxin, Type A, Lower Dose 1
  botulinum toxin, Type A: topical liniment
- ET-01 1100U: botulinum toxin, Type A, Higher Dose 2
  botulinum toxin, Type A: topical liniment
Arm/Group | Vehicle | ET-01 345U | ET-01 1100U
Number analyzed (Participants) | 23 | 30 | 19
Number analyzed (Observations) | 68 | 88 | 57
Observations | 4 | 6 | 8

ADVERSE EVENTS:
Time Frame: 26 weeks
Arm/Group | Vehicle | ET-01 345U | ET-01 1100U
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/30 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/30 | 0/20
Other Adverse Events (participants affected / at risk) | 13/25 | 4/30 | 5/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vehicle (N=25) | ET-01 345U (N=30) | ET-01 1100U (N=20)
Application site pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Blepharitis (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Cough (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Cystitis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Ear infection (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Endodontic procedure (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Endometrial ablation (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (General disorders) | 2 (2) | 0 (0) | 0 (0)
Hordeolum (Eye disorders) | 4 (4) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Mammoplasty (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Nail dystrophy (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 4 (4)
Nausea (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0)
Rhinitis allergic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0)
Skin discolouration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Thyroiditis subacute (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Study Results are considered Confidential Information that may not be published or disclosed without Sponsor's written consent for a period of five (5) years after completion of the Study.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-06): https://cdn.clinicaltrials.gov/large-docs/93/NCT03839693/Prot_SAP_000.pdf